CLINICAL TRIAL: NCT06007651
Title: A Phase 1, Multicenter, Randomized, Placebo-Controlled, Double-Blind Trial of LY3885125 to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of a Single Ascending Dose in Participants With Dyslipidemia and Repeat-Doses in Participants With NAFLD
Brief Title: A Study of LY3885125 in Participants With Dyslipidemia or Non-Alcoholic Fatty Liver Disease (NAFLD)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Participants were not dosed in Part B as per the protocol, the patient population will be refined and new outcome measures will be applied in a separate study.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 18769; J4N-MC-YFAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-08-18; First posted 2023-08-23 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Dyslipidemias; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Dyslipidemias; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- LY3885125 (Part A) (Experimental): Single ascending doses of LY3885125 administered subcutaneously (SC)
  Interventions: Drug: LY3885125
- Placebo (Part A) (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo
- LY3885125 (Part B) (Experimental): Repeat doses of LY3885125 administered SC
  Interventions: Drug: LY3885125
- Placebo (Part B) (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3885125 — Administered SC
  Arms: LY3885125 (Part A); LY3885125 (Part B)
Drug: Placebo — Administered SC
  Arms: Placebo (Part A); Placebo (Part B)

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3885125 after administration of single ascending doses in participants with dyslipidemia (part A) and multiple doses in participants with non-alcoholic fatty liver disease (part B). Blood tests will be performed to check how much LY3885125 gets into the bloodstream and how long it takes the body to eliminate it.

The study will last up to approximately 49 weeks for part A and 62 weeks for part B, for a total of approximately 111 weeks.

ELIGIBILITY:
Inclusion Criteria:

Parts A & B

* Males, or females of not of childbearing potential,
* On a stable diet for the 3 months prior to randomization and willing to continue the same stable diet during the study.

Part A

* Dyslipidemia with the following fasted blood levels at screening: 150 mg/dL ≤ triglycerides <500 mg/dL, AND LDL-cholesterol ≥100 mg/dL,
* Body mass index (BMI) in range of 18.5 to 45.0 kg/m2. Part B
* NAFLD with liver fat content ≥8% as determined by magnetic resonance imaging proton density fat fraction (MRI-PDFF),
* BMI in range of 27 to 45.0 kg/m2

Exclusion Criteria:

Parts A & B

* History or presence of medical illness including, but not limited to, any cardiovascular, thromboembolism or bleeding disorder, hepatic, respiratory, hematological, endocrine, immune, psychiatric, or neurological disease, convulsions, or any clinically significant laboratory abnormality that, in the judgment of the Investigator, indicate a medical problem that would preclude study participation,
* Uncontrolled hypertension with a resting blood pressure ≥ 160 mmHg systolic or ≥ 100 mmHg diastolic at visit 1,
* Alanine transaminase (ALT) or aspartate aminotransferase (AST) >3.0 × ULN for the reference range,
* Alkaline phosphatase (ALP) >1.5 × ULN for the reference range,
* Total bilirubin (TBL) >1.5 × ULN for the reference range,
* Taken drugs associated with hepatic steatosis (e.g., amiodarone, valproic acid, methotrexate, tamoxifen) for more than 2 weeks in the 3 months prior to screening visit,
* Type 1 diabetes mellitus (T1DM) or any other type of diabetes mellitus other than T2DM,
* Poorly controlled T2DM with glycated hemoglobin (HbA1c) of >9.0%,
* Treatment with GLP-1 RA and GIP/GLP-1 RA and approved or experimental agents that target PCSK9 within 9 months prior to screening visit.

Part B

* Evidence of other forms of chronic liver disease,
* Initiated treatment with, or changed dose of, medications that may cause significant weight gain or weight loss, within 3 months prior to the screening visit,
* Have a self-reported change in body weight >5 kg (11 pounds) within 3 months prior to screening visit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Part A: Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to 49 weeks (Part A)
  Part A: A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module
Part B: Number of Participants with One or More SAEs Considered by the Investigator to be Related to Study Drug Administration | Baseline up to 62 weeks (Part B)
  Part B: A summary of SAEs and other non-serious AEs, regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Part A & B: Pharmacokinetics (PK): Area Under the Plasma Concentration Versus Time Curve (AUC) of LY3885125 | Baseline up to 49 weeks (Part A) and Baseline up to 62 weeks (Part B)
  Part A & B: PK: AUC of LY3885125
Part A & B: PK: Maximum Observed Plasma Concentration (Cmax) of LY3885125 | Baseline up to 49 weeks (Part A) and Baseline up to 62 weeks (Part B)
  Part A & B: PK: Cmax of LY3885125
Part A & B: PK: Time of Maximum Observed Concentration (Tmax) of LY3885125 | Baseline up to 49 weeks (Part A) and Baseline up to 62 weeks (Part B)
  Part A & B: PK: Tmax of LY3885125
Part A & B: Pharmacodynamics (PD): Change From Baseline in Proprotein Convertase Subtilisin/Kexin type 9 (PCSK9) | Baseline up to 49 weeks (Part A) and Baseline up to 62 weeks (Part B)
  Part A & B: PD: Change From Baseline in PCSK9
Part A & B: PD: Change From Baseline in apolipoprotein B (ApoB) | Baseline up to 49 weeks (Part A) and Baseline up to 62 weeks (Part B)
  Part A & B: PD: Change From Baseline in ApoB
Part B only: PD: Change of Liver Fat Content From Baseline by Magnetic Resonance Imaging Proton Density Fat Fraction (MRI-PDFF) | Baseline up to 62 weeks (Part B)
  Part B only: PD: Change of Liver Fat Content From Baseline by MRI-PDFF

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Worldwide Clinical Trials, Inc., San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No